CLINICAL TRIAL: NCT05270564
Title: Post-operative Drainage After Pancreaticoduodenectomy: A Randomized Controlled Trial of Patients With Intermediate and Low Risk for Pancreatic Fistula
Brief Title: Post-operative Drainage After Pancreaticoduodenectomy
Acronym: Drain 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Bergthor Björnsson, Associate Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Drain_1
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (Active Comparator): Surgical drains used as routine
  Interventions: Procedure: Drain
- No drain (Experimental): No surgical drain used
  Interventions: Procedure: No drain

INTERVENTIONS:
Procedure: Drain — Surgical drains are placed as a standard of care (control arm) or not (experimental arm)
  Arms: Drain
Procedure: No drain — Surgical drains are placed as a standard of care (control arm) or not (experimental arm)
  Arms: No drain

SUMMARY:
The study compares regular use of surgical drains and no use of surgical drains in patients subjected to pancreaticoduodenectomy with expected low to intermediate risk for post operative pancreatic fistula.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy of both sexes
* Patients with predicted risk score of 10 or less of pancreatic fistula
* Written informed consent
* Expected survival time > 6 months

Exclusion Criteria:

* Patients with predicted high risk of fistula with a risk score above 10
* Patients with intraabdominal abscess or infection
* ASA score > 3
* Pregnancy
* Expected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall morbidity rate | 90 days post operatively
  Post operative morbidity

SECONDARY OUTCOMES:
Mortality rate (in-hospital, 30 and 90 days) | 90 days post operatively
Severe morbidity rate as classified by Clavien-Dindo >3 | 90 days post operatively
Fistula rate according to ISGPF | 90 days post operatively
Intraabdominal abscess rate | 90 days post operatively
Wound infection rate | 90 days post operatively
Delayed gastric emptying according to ISGPF | 90 days post operatively
Postpancreatectomy bleeding according to ISGPF | 90 days post operatively
Need of interventional radiology | 90 days post operatively
Need for reoperation | 90 days post operatively
Hospital stay | 90 days post operatively
Readmission rate | 90 days post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Bergthor Björnsson, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Linkoping University Hospital, Linköping
  - Skanes University Hospital, Lund

IPD SHARING:
Plan to Share IPD: No